CLINICAL TRIAL: NCT01570699
Title: COMT Val158Met Polymorphism in Opiate-using Subjects Without Lifetime Opiate Dependence
Brief Title: Variation of COMT Val158Met Polymorphism Between COM-ON Patients and METHADOSE Patients
Acronym: COM-ON
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC10 073; 2011-A00623-38 (Other: IDRCB)
Record Dates: First submitted 2012-02-02; First posted 2012-04-04 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Opioid-related Disorders; Opiate Dependence; Opiate Addiction; Opiate Abuse
Keywords: Cross-sectional observational study; COMT polymorphism; Opiate-users; Opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will compare polymorphism COMT between COM-ON patients and METHADOSE patients. Samples may be blood sample or salivary sample.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2: patients included in METHADOSE study: includes opiate-dependent patients substituted by methadone
  Interventions: Genetic: COMT polymorphism
- 1: opiate-non dependent patients: Will be included in the COM ON study subjects who have consumed illicit opiates (heroin, methadone, buprenorphine or morphine) more than 10 times in their life, without ever having the DSM-IV criteria for opiate dependence or abuse
  Interventions: Genetic: COMT polymorphism

INTERVENTIONS:
Genetic: COMT polymorphism — The COMT enzyme enables the degradation of brain monoamines such as Dopamine and is encoded by a single gene for which several polymorphisms are known, including the Val158Met polymorphism which has been widely studied in various psychiatric disorders including addictions, as well as in impulsivity

SUMMARY:
The main objective is to compare the genotypes of the COMT Val158Met polymorphism between opiate-users and opiate-dependent subjects. The secondary objective is to constitute a sample of opiate-users without any lifetime opiate dependence.

DETAILED DESCRIPTION:
The COMT enzyme enables the degradation of brain monoamines such as Dopamine and is encoded by a single gene for which several polymorphisms are known, including the Val158Met polymorphism which has been widely studied in various psychiatric disorders, including addictions, as well as in impulsivity. In most studies it is the Val allele which is found to be associated with addictive behaviors. The study METHADOSE, which began in 2009, includes opiate-dependent patients substituted by methadone. The preliminary analysis of this study shows a genotype distribution different from that of general population samples, with a greater prevalence of Val / Val and Val / Met genotypes. Will be included in the COM ON study subjects who have consumed illicit opiates (heroin, methadone, buprenorphine or morphine) more than 10 times in their life, without ever having the DSM-IV criteria for opiate dependence or abuse. The study will compare, by means of saliva samples, Val / Val and Val / Met genotypes between the subjects recruited in COM ON and those recruited in METHADOSE. Will also be included auto-questionnaires to identify psychological factors that may constitute risk or protective factors vis-à-vis the development of dependence.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Caucasian patients
* Clinical diagnosis of lifetime opiate-using disorder (consumption over 10 times of illicit opiates (heroin, buprenorphine, methadone or morphine))
* Not lifetime history of opioid dependence (DSMIV)
* Patients with health insurance coverage
* Patient was treated with opioids analgesics to alleviate 2 or 3 in their lives

Exclusion Criteria:

* Non-Caucasian patients
* Patients who cannot give their consent and/or who refuse the collection of genetic data
* Patients with no health insurance coverage

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who have consumed illicit opiates (heroin, methadone, buprenorphine or morphine) more than 10 times in their life, without ever having the DSM-IV criteria for opiate dependence or abuse
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with each COMT genotype (Val/Val, Val/Met and Met/Met) in the opiate-users' group and in the opiate-dependent subjects' group | Day 0

SECONDARY OUTCOMES:
Score on the M.I.N.I. (Mini-International Neuropsychiatric Interview) on the day of the inclusion | Day 0
Score on the BIS (Barratt Impulsivity Scale) on the day of the inclusion | Day 0
Score on the TCI (Cloninger's Temperament and Character Inventory) on the day of the inclusion | Day 0
Score on the WURS (Wender Utah Rating Scale) on the day of the inclusion | Day 0
Score on the ASRS(Self-Report Scale) on the day of the inclusion | Day 0
Score on the MOPS (Measure Of Parental Style) on the day of the inclusion | Day 0
Score on the Questionnaire of family breakdowns on the day of the inclusion | Day 0
Score on the CD-RISC (Connor-Davidson Resilience scale) on the day of the inclusion | Day 0
Score on the CTQ (Childhood trauma questionnaire) on the day of the inclusion | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Florence VORSPAN, MD, MSC, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Espace Murger, Consultation toxicomanie, Fernand-Widal Hospital (AP-HP), Paris, Île-de-France Region, France